CLINICAL TRIAL: NCT00318240
Title: Feasibility Study for Locally Recurrent Prostate Cancer Treatment Following Radiation Failure With High Intensity Focused Ultrasound (HIFU)
Brief Title: Prostate Cancer Treatment Following Radiation Failure With High Intensity Focused Ultrasound (HIFU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-05-877; 11936
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
Keywords: High Intensity Focused Ultrasound; Men; Locally recurrent prostate cancer.
MeSH Terms: conditions — Prostatic Neoplasms; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): High Intensity Focused
  Interventions: Device: High Intensity Focused Ultrasound

INTERVENTIONS:
Device: High Intensity Focused Ultrasound — Treatment of Radiation failure in Prostate Cancer
  Other Names: HIFU

SUMMARY:
This is a feasibility study to determine safety and the ability of HIFU (High Intensity Focused Ultrasound)to selectively destroy prostate cancer tissue in men who demonstrate local recurrence of prostate cancer following radiation treatment.

DETAILED DESCRIPTION:
This is a feasibility study to determine the safety and the ability of HIFU (High Intensity Focused Ultrasound)to selectively destroy prostate cancer tissue in men who demonstrate local recurrence of prostate cancer following radiation treatment. All participants will receive treatment with HIFU and be monitored closely for recurrence of disease (if any),quality of life and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* · Male patients with an initial presentation of organ confined recurrent prostate cancer (clinical Stages T1 and T2 only) who have been treated with external beam radiation therapy or brachytherapy and subsequently has biopsy-proven local recurrence.

  * Age > 40 years through <80 years.
  * Anesthesia Surgical Assignment (ASA) categories I, II or III only.
  * Negative radionuclide bone scan within 3 months prior to HIFU treatment to rule out the possibility of metastases.
  * PSA levels >0.5ng/ml and <10ng/ml.
  * Pre-radiation Gleason score < 8
  * Clearly imageable prostate on TRUS
  * Written informed consent.

Exclusion Criteria:

* · T3 or T4 prostate cancer.

  * Age <40 years. or >80 years.
  * ASA of IV and higher.
  * Gleason score>8.
  * PSA <0.5ng/ml or >10ng/ml.
  * Prostate size > 40 grams as determined by transrectal ultrasound
  * Large calcification in the area to be treated (>5mm).
  * Bleeding disorder as determined by abnormal prothrombin time (INR)and partial thromboplastin time (PTT).
  * Patient on Coumadin or any other anticoagulant, unless their anticoagulation can be temporarily reversed or stopped.
  * Urinary tract infection unless treated satisfactorily by antibiotics and documented by a sterile urine culture.
  * Interest in future fertility.
  * History of allergy to latex.
  * Inability to visualize the prostatic tissue adequately on transrectal ultrasound imaging.
  * Currently on hormonal therapy for prostate cancer (patients can be enrolled if they come off hormone therapy for 3 months).
  * History of treatment for prostate cancer, other than brachytherapy or external beam radiation.
  * History of TURP, thermotherapy or urethral stent.
  * History of any major rectal surgery.
  * History of inflammatory bowel disease.
  * History of urinary bladder neck contracture.
  * History of any other malignancy other than skin cancer.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of HIFU in men with local recurrent prostate cancer following radiation therapy. | ongoing

SECONDARY OUTCOMES:
Destruction of prostate cancer tissue. | ongoing
Safety of repeating procedure in patients who do not respond adequately. | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Joseph Chin, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada